CLINICAL TRIAL: NCT05132634
Title: Evaluation of the Effect of Hand Massage in Prevention of Pressure Wound
Brief Title: The Effect of Massage in Preventing Pressure Wound Development
Acronym: PW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Esra Ozkan, Lecturer, Giresun University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Giresun University
Record Dates: First submitted 2021-10-27; First posted 2021-11-24 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Pressure Injury
Keywords: Massage; Nursing Care; Pressure Ulcer; Therapeutic touch
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Paralel Assignment randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms (Experimental): Experimental Group:
  Braden Risk Assessment Scale was completed on the first day of admission to the Intensive Care Unit and every morning in the morning.
  Since the care hours were between 08:00_10:00 in the morning and 20:00-22:00 at night, classical hand massage was applied to the patient by the researcher between the time zones specified daily.
  It was followed up with the Pressure Wound Staging Form.
  Control Group:
  The Braden Risk Assessment Scale was completed on the first day of admission to the Intensive Care Unit and every morning in the morning.
  It was followed up with the Pressure Wound Staging Form.
  Interventions: Other: Hand Massage

INTERVENTIONS:
Other: Hand Massage — Like a massage, the superficial kneading technique which is included in the Swedish massage technique will be applied in a way to create a slight pressure on the patient, and it will be terminated again with the effleurage technique. The procedure was concluded in a way that each massage technique was applied and the massage was for a total of 15-20 minutes.

SUMMARY:
Pressure Wound (PW) is a chronic wound that develops in soft tissue as a result of the capillary end pressure which rising above 32 mmHg. It is the most common complication with 31% annual incidence after spinal cord injuries. Pressure wound is considered as malpractice for nursing practices. It decreases the quality of life of the elderly and patients with mobility restrictions and prolongs the length of hospital stay. Complication development risk and cost are high. Factors affecting wound opening include the amount of pressure, duration, moisture, friction, nutrition, age, weight, hemoglobin value, chronic diseases. The development of preventive actions, protocol and standard in pressure wound planning of care is among the main goals of nursing care. The research will be carried out to evaluate the effect of hand massage in preventing pressure injuries. Patient with a high risk of developing pressure wound will constitute the experimental and control group of our study. Standard nursing care applied to the control group; unlike the control group hand massage will be applied to the experiment group.when the sample group determined in both the experimental and control groups is reached the study will be terminated. The pressure wound in both groups will be compared statistically and the effectiveness of hand massage in reducing the pressure wound will be determined.

H0 :The applied classical hand massage has no effect on the formation of pressure wound.

H1: The applied classical hand massage has effect on the formation of pressure wound.

DETAILED DESCRIPTION:
Background: According to the National Pressure Ulcer Association Panel (NPUAP) data, the incidence of pressure wounds (PW) in acute care units varies between 0.4-38%, in long-term care units 2.2-23.9%. While it is stated that more than 700,000 patients develop PW each year in the UK and 180,000 of them start in the hospital, PW is a significant health burden affecting more than 2.5 million adults per year in the United States (USA) and will affect the growing elderly population in the future. According to the National Health Service (NHS), it is claimed that the daily cost of treatment applied in the treatment of PW is more than 3.8 million. European Pressure Ulcer Association Panel (EPUAP) according to, PW is defined as localized skin/subcutaneous tissue damage, usually occurring on bone prominences, caused by additional factors together with pressure or shearing. It is said that hand massage is effective in preventing the development of PW; when the literature results are examined, it has been determined that there are insufficient studies at the level of evidence to measure the effectiveness of massage applications or hand massage. Therefore, our study, it was aimed to evaluate the effect of classical hand massage on the prevention of PW.

Method: A total of 60 patients over the age of 18 who were hospitalized in the intensive care unit of the hospital with undeveloped PW and who had not undergone surgery were randomly assigned to the experimental and control groups. The patients included in the experimental group were massaged twice a day, in the morning and evening, together with nursing care, for 15-20 minutes. Admitted to the control group. only nursing care was applied to the basta. Due to the lack of a clear time for PW development in the literature, patients; In the hospital where the research was conducted, patients were followed up for 12 days, since the average duration of opening RF was 12 days in 2019-2020. Patients who were opened BY were followed up until the day they were opened.

ELIGIBILITY:
Inclusion Criteria:

* Being in the intensive care unit, being 18 years or older,
* Braden Risk Assessment Scale score 12 and below,
* Patients whose position change is within the scope of the physician's request (patients whose position change is not restricted such as spinal cord injury, orthopedic surgery),
* Conscious patients willing to participate in the study or obtaining permission from family members in the unconscious.

Exclusion Criteria:

* Having a Braden Risk Assesment Scale (BRAS) score of 12 and above,
* Staying in the intensive care unit for less than five days, Pressure wound Stage 1 and above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | 6 months
  The form (22, 52) developed by the researcher in line with the literature, the patient group (experimental, control), age, gender, presence of chronic disease, current chronic disease, physical evaluation (height, weight, body mass index), hospitalization cause/diagnosis, fluid intake and nutritional status, pressure ulcer formation status, number, region, day and time of occurrence, Braden Risk Assessment Scale score. Of these statements, 11 are for all patients in both groups with and without pressure ulcers, and four for patients who only develop pressure ulcers. The data in this form were collected through observation and obtained from the nurse observation form.Sociodemographic characteristics of the patients will be measured.

OTHER OUTCOMES:
Pressure Wound Staging Form | 6 months
  Staging was performed according to the National Pressure Ulcer Panel Pressure Ulcer Injuries Staging System Stage 1: Skin integrity is intact. There is redness that does not fade with pressure on the skin in other areas, mostly bone protrusions. The wound site may be painful, hard, soft, warmer or colder than the surrounding tissues.
Experimental and Control Group Follow-up Form | 6 months
  It was created by the researcher, using the literature information, in order to follow the patient's laboratory values and the skin in risky areas in terms of the formation of pressure wound. It was recorded for the patients included in the experimental group in the daily experimental group follow-up form by being evaluated every day and at each position hour in terms of A clear disc was used during skin diagnosis to evaluate non-whitening erythema more objectively. When RA developed in the areas under observation, the follow-up of the area with pressure sores was terminated. Since the laboratory values of the patients were checked weekly in the unit where the study was conducted, albumin and hemoglobin values were obtained from the patient file. Laboratory values were evaluated by considering the values in the reference range of the hospital where the research was conducted

CONTACTS AND LOCATIONS:
Overall Officials: Esra Özkan, Lecturer, Principal Investigator — Giresun University Health Servives Vocational School
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://www.sciencedirect.com/science/article/pii/S0020748921001619 — https://doi.org/10.1016/j.ijnurstu.2021.104014